CLINICAL TRIAL: NCT04671550
Title: Glaucoma and Driving Licence: How to Identify Patients at Risk of Having it Revoked
Brief Title: The Value of Visual Field Examination in Driving Licence.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Simone Donati, Associate Professor, Università degli Studi dell'Insubria
Other Study IDs: 2020/Glaucoma
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Glaucoma Eye
Keywords: visual field; driving licence; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: questionnaire — Questionnaire on "Driving performances and Visual Field"

SUMMARY:
The aim of the study is to identify clinical criteria, easily achievable with patient's follow-up tests, which can identify individuals at increased risk of being unfit to drive. Only they, then, will be directed to further investigations. These clinical standards should also be suitable for implementing or substituting the current law's criteria, after appropriate additional studies, so that the law can be based on the clinic.

DETAILED DESCRIPTION:
In this observational study, the investigators recruite patients referred at the Glaucoma Service of the Ophthalmologic Clinic of the ASST Sette Laghi University Hospital in Varese.

All the patients enrolled in the study require a reliable (less than 15% of false positive or false negative and no more than 33% of loss of fixation) visual field examination (Humphrey SITA 24-2 or 30-2 SITA Standard) performed in the previous six months.

All patients undergo a full ophthalmologic examination and verbally submitted a questionnaire designed by the authors of the paper (LL, SD, MD).

The examination included Visual Acuity, refraction, slit lamp bio-microscospy, Goldmann's applanation tonometry, gonioscopy with four mirror lens, OCT RNFL and GCL imaging if necessary and re-evaluation of target IOP.

The investigators use the two monocular visual fields to build an Integrated Visual Field which, according to D.P. Crabb papers, is an efficient surrogate to the Binocular Esterman Visual Field Test (EVFT). In short, each point in each monocular field is compared to its equivalent in the other eye, and the data, from the eye with the best sensitivity, are used. Locations are dichotomized into groups with sensitivity > 10 dB and < 10 dB, representing whether a patient would see or miss a point in the Esterman test, respectively. To match even better the IVF with the EVFT, 8 points of the inner 20° of the IVF were excluded since they have no direct equivalent in the EVFT.

ELIGIBILITY:
Inclusion Criteria:

* subjects above 18 years of age
* clear diagnosis of Glaucoma (of any type)
* to show a reliable (less than 15% of false positive or false negative and no more than 33% of loss of fixation) visual field examination (Humphrey SITA 24-2 or 30-2 SITA Standard) performed in the previous six months.

Exclusion Criteria:

* other ocular conditions that could affect the visual field (i.e. cataract or macular degeneration).
* patients that underwent a 10-2 test since it does not allow the composition of the Integrated Visual Field.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators recruite patients referred at the Glaucoma Service of the Ophthalmologic Clinic of the ASST Sette Laghi University Hospital in Varese
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Visual Field quality by combining two parameters obtained by Computerized Visual Field Examination: number of missed points within the central 20° visual field and average Sensitivity (AS) of all the 60 points of the 24-2 grid | Baseline
  The Visual Field quality will be evaluated by considering two variables: Number of missed points within the central 20° visual field (expressed in number) and average Sensitivity (AS) of all the 60 points of the 24-2 grid (expressed in decibel, dB)

SECONDARY OUTCOMES:
Creation of a Integrated Visual Field of both eyes | Baseline
  Composition of the Visual Fields of both eyes of the same subject obtained by the Cmputerized Visual Field by integrating average sensitivity expressed in decibel (dB) and the missed points expressed in pure numbers.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided